CLINICAL TRIAL: NCT03462147
Title: The Efficacy of Spinal Cord Stimulation in Patients With a Failed Back Surgery Syndrome.
Brief Title: Efficacy of Spinal Cord Stimulation in Patients With a Failed Back Surgery Syndrome.
Acronym: HDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Dieter Mesotten, MD, Ziekenhuis Oost-Limburg
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Device Feasibility
Other Study IDs: HDS study
Record Dates: First submitted 2018-03-01; First posted 2018-03-12 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Back Pain; Spinal Cord Stimulation
MeSH Terms: conditions — Back Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Intervention Model Description: We wish to compare different stimulation modes within a patient population in which an epidural electrode for FBSS has been implanted, in order to evaluate the effectiveness. We will evaluate the modality "high-density", conventional stimulation and sham stimulation in the same patient. This can be easily adjusted by reprogramming the implanted battery.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHAM (Sham Comparator): No stimulation will be given
  Interventions: Device: Spinal cord stimulation
- High Density Stimulation (Experimental): New way of spinal cord stimulation
  Interventions: Device: Spinal cord stimulation
- Conventional stimulation (Active Comparator): the most used stimulation of the spinal cord
  Interventions: Device: Spinal cord stimulation

INTERVENTIONS:
Device: Spinal cord stimulation — Spinal cord stimulation will be given according to the arms of the group (no stimulation, high density stimulation of conventional stimulation)

SUMMARY:
When patients suffer from chronic pain after multiple back surgeries, this is denominated as the 'failed back surgery syndrome'. A possible treatment for these patients is spinal cord stimulation. This is an invasive treatment where no other treatment options (medication, minimal invasive treaments) can offer progress to the patients' health status. In spinal cord stimulation, an electrode will be placed at the spinal cord under local anaesthesia whereas via a battery a painless electrical stimulation will arise. Clinical research have demonstrated that a new way of spinal cord stimulation can improve back and leg pain significantly. This will lead to a better quality of life for the patients and a decreased use of medications. In Ziekenhuis Oost-Limburg, different manners of spinal cord stimulation will be compared to each other.

DETAILED DESCRIPTION:
The patients in our pain centre are implanted with Medtronic material. This material cannot deliver the 10kHz frequency but can deliver up to 5000 Hz (hereinafter referred to as high density stimulation). This also delivers high energy to the spinal cord without palpable paresthesia, with a beneficial effect on the pain.

We wish to include patients who, in accordance with Belgian regulations, have undergone a normal evaluation period with an external battery and who have subsequently had a definitive system implanted. The implant procedure, evaluation period and the material used are identical to patients outside the study context.

We wish to compare different stimulation modes within a patient population in which an epidural electrode for failed back surgery syndrome (FBSS) has been implanted, in order to evaluate the effectiveness. We will evaluate the modality "high-density", conventional stimulation and sham stimulation in the same patient. This can be easily adjusted by reprogramming the implanted battery. For this study we want to use a relatively new study design, namely: single case design (N-of-1 trial). In this, many variables will be evaluated with a limited number of study subjects in order to determine an effect. We want to investigate to what extent the patient experiences the different stimulation modes and to what extent he can compare or prefer these stimulation modes. The stimulation that the patient prefers as most pleasant can be continued afterwards. If the patient does not experience pain reduction during a certain stimulation mode, he can always fall back on his own pain medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an implanted neurostimulation system met een FBSS met geïmplanteerd

Exclusion Criteria:

* no knowledge of the Dutch language
* Addicted to drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of pain | 28 days
  Pain will be evaluated in the different groups according to a pain scale varying from 1 to 11 with 0 no pain and 11 a lot of pain

SECONDARY OUTCOMES:
Need of medication | 28 days
  The difference in medication in the different groups will be assessed using a questionnaire
Quality of life and functional outcome | 28 days
  Quality of life will be assessed according to a questionnaire
Quality of sleep | 28 days
  Quality of sleep will be assessed according to a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Martine Puylaert, MD PhD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium

REFERENCES:
- [Derived] O'Connell NE, Ferraro MC, Gibson W, Rice AS, Vase L, Coyle D, Eccleston C. Implanted spinal neuromodulation interventions for chronic pain in adults. Cochrane Database Syst Rev. 2021 Dec 2;12(12):CD013756. doi: 10.1002/14651858.CD013756.pub2. PMID 34854473